CLINICAL TRIAL: NCT00066404
Title: A Phase I Clinical Trial of Intrapleural Adenoviral-Mediated Interferon-beta (IFN-ß) Gene Transfer for Pleural Malignancies
Brief Title: Intrapleural BG00001 in Treating Patients With Malignant Pleural Mesothelioma or Malignant Pleural Effusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000315899; UPCC-01502
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cancer
Keywords: advanced malignant mesothelioma; male breast cancer; localized malignant mesothelioma; recurrent bladder cancer; recurrent renal cell cancer; recurrent urethral cancer; recurrent breast cancer; recurrent penile cancer; recurrent prostate cancer; recurrent anal cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent gastric cancer; recurrent pancreatic cancer; recurrent rectal cancer; recurrent gastrointestinal carcinoid tumor; recurrent small intestine cancer; recurrent gallbladder cancer; recurrent extrahepatic bile duct cancer; recurrent adult primary liver cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; recurrent thymoma and thymic carcinoma; recurrent melanoma; recurrent malignant mesothelioma; recurrent malignant testicular germ cell tumor; recurrent cervical cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; recurrent vulvar cancer; recurrent vaginal cancer; recurrent gestational trophoblastic tumor; recurrent endometrial carcinoma; recurrent ovarian germ cell tumor; malignant pleural effusion
MeSH Terms: conditions — Neoplasms; Breast Neoplasms, Male; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Urethral Neoplasms; Breast Neoplasms; Penile Neoplasms; Prostatic Neoplasms; Anus Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thymoma; Melanoma; Mesothelioma, Malignant; Testicular Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Gestational Trophoblastic Disease; Endometrial Neoplasms; Pleural Effusion, Malignant

INTERVENTIONS:
Biological: recombinant adenovirus-hIFN-beta

SUMMARY:
RATIONALE: Using BG00001 to insert the gene for interferon-beta into a person's pleural cavity may improve the body's ability to fight cancer.

PURPOSE: Phase I trial to study the effectiveness of intrapleural BG00001 in treating patients who have malignant pleural mesothelioma or malignant pleural effusions.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of intrapleural BG00001 in patients with malignant pleural mesothelioma or malignant pleural effusions.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the success of gene transfer/interferon beta gene expression in patients treated with this drug.
* Determine systemic and intrapleural cytokine responses and cellular and humoral immune response in patients treated with this drug.
* Determine, preliminarily, tumor response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive BG00001 via an intrapleural catheter on day 1.

Cohorts of 3-6 patients receive escalating doses of BG00001 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

Patients are followed weekly for 1 month, biweekly for 1 month, monthly for 4 months, and then every 6 months for 15 years.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically or cytologically confirmed diagnoses:

  * Malignant pleural mesothelioma
  * Metastatic malignancy to the pleural space

    * Originating from 1 of the following sites:

      * Lung
      * Breast
      * Gastrointestinal organs
      * Genitourinary organs
      * Malignant melanoma
    * Failed prior standard therapy comprising chemotherapy, radiotherapy, and/or hormonal therapy
* Measurable or evaluable disease
* Pleural space involved with tumor accessible for pleural catheter insertion
* No malignant pleural effusions secondary to lymphoma or sarcoma
* No rapidly re-accumulating, symptomatic pleural effusions after thoracentesis or pleural catheter insertion that require immediate mechanical or chemical pleurodesis
* No known brain metastases

  * Previously treated brain metastases with no evidence of active growth are allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit at least 30% (transfusion allowed)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* PT and PTT no greater than 1.5 times normal
* No end-stage liver disease
* No chronic active hepatitis B (hepatitis B surface antigen negative)

Renal

* Creatinine no greater than 2.0 mg/dL
* No end-stage renal disease

Cardiovascular

* No unstable angina

Pulmonary

* FEV_1 greater than 50% of predicted (post-pleural drainage)
* No severe oxygen-dependent chronic obstructive pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No documented immunodeficiency
* No other malignancy within the past 5 years except nonmelanoma skin cancer or successfully treated localized malignancy of the bladder or prostate gland with no evidence of active disease
* No other life-threatening illness
* No known hypersensitivity to any component of study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy
* No prior bone marrow transplantation, including stem cells
* No immunological drugs during and for at least 2 months after study therapy

Chemotherapy

* See Disease Characteristics
* No chemotherapy during and for at least 2 months after study therapy

Endocrine therapy

* See Disease Characteristics
* Concurrent hormonal therapy allowed if maintained at dose received prior to study entry
* No concurrent steroids

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No radiotherapy during and for at least 2 months after study therapy

Surgery

* At least 2 weeks since prior surgery

Other

* More than 4 weeks since prior cytotoxic agents
* No concurrent immunosuppressives or medication that can directly or indirectly suppress the immune system
* No other concurrent experimental therapies for pleural cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Sterman, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Sterman DH, Recio A, Haas AR, Vachani A, Katz SI, Gillespie CT, Cheng G, Sun J, Moon E, Pereira L, Wang X, Heitjan DF, Litzky L, June CH, Vonderheide RH, Carroll RG, Albelda SM. A phase I trial of repeated intrapleural adenoviral-mediated interferon-beta gene transfer for mesothelioma and metastatic pleural effusions. Mol Ther. 2010 Apr;18(4):852-60. doi: 10.1038/mt.2009.309. Epub 2010 Jan 12. PMID 20068553